CLINICAL TRIAL: NCT04833556
Title: Clinical Characteristics and Perioperative Outcomes of Postpartum Hemorrhage in Patients Undergoing Cesarean Delivery
Brief Title: Perioperative Outcomes of Postpartum Hemorrhage in Patients Undergoing Cesarean Delivery
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Other Study IDs: 005/2564 (IRB4); 161/2021 (Registry Identifier: Siriraj Institutional Review Board COA number)
Record Dates: First submitted 2021-04-01; First posted 2021-04-06 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Cesarean Section Complications; Postpartum Hemorrhage; Anesthesia Complication; Blood Transfusion Complication; Uterine Atony With Hemorrhage
Keywords: Cesarean section; Postpartum haemorrhage; Anesthesia complication; Blood transfusion; Intensive care unit admission
MeSH Terms: conditions — Postpartum Hemorrhage; Transfusion Reaction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Postpartum haemorrhage: Patients undergoing cesarean delivery with postpartum haemorrhage (blood loss more than or equal to 1,000 ml.)

SUMMARY:
Postpartum haemorrhage is the common cause of maternal death worldwide. The primary purpose of this study is to identify the maternal outcomes after PPH. The highlighted outcome is the anesthetic management including rate of blood transfusion and incidence of patient experiencing massive blood transfusion. The secondary purposes of this study are amount of blood loss, causes of PPH and other outcomes that related to PPH such as the rate of hysterectomy and postoperative outcome eg. congestive heart failure, acute kidney injury and TRALI etc. Additionally, incidence of PPH will be studied. Data collection will be made to identify the cause of PPH, anesthetic techniques that may related to the amount of hemorrhage, medical treatment for PPH and neonatal outcomes. We also aim to obtain the rate of ICU admission and revealed the factors involving the ICU admission in PPH patients underwent cesarean delivery.

DETAILED DESCRIPTION:
Postpartum hemorrhage (PPH) is the common cause of maternal death worldwide. It is interesting to note that PPH is the most common cause of death in developing country. Additionally, PPH is the common cause of maternal cardiac arrest. PPH defined as the amount of bleeding more than or equal to 500 ml after vaginal delivery and bleeding of more than or equal to 1,000 ml after cesarean delivery. The rate of PPH regardless any route of delivery was 2.9-3.2%. Rate of PPH in patients undergoing cesarean delivery was approximately 0.6% - 3.1%.

The difference in anesthetic techniques influence the rate of postpartum hemorrhage. Numerous studies showed the association between general anesthesia and postpartum hemorrhage in patient undergoing cesarean delivery. The outcome showed the odds of PPH in women who had cesarean delivery with general anesthesia were 8.15 times higher (95% CI 6.43-10.33) than for those who had CS with epidural anesthesia. Likewise, systematic review and meta-analysis revealed general anesthesia associated with higher amount of blood loss, but not the transfusion rate comparing with regional anesthesia. The decreasing of myometrial uterine tone from the usage of inhalational agents (halothane, enflurane, isofurane, sevoflurane, and desflurane) from general anesthesia explains this consequence.

Guidelines recommended the management of PPH after cesarean delivery were launched. World Health Organization (WHO) recommendation reported both surgical together with medical management (non-surgical) in patients with PPH, which published in the year 2012. The major role of anesthesiologists involving in treatment of PPH is medical treatment and blood and blood component administration. The novel medical treatment of PPH has been described in several literatures including the usage of tranexamic acid and fibrinogen concentrate. The World Maternal Antifibrinolytic trial (WOMAN trial) is the large-sample size randomized controlled trial publishing in the Lancet in the year 2017. WOMAN trial revealed the administration of tranexamic acid in patients with PPH after vaginal or cesarean delivery significantly reduced blood loss and decreased maternal mortality rate from bleeding. Likewise, Cochrane database systematic review concluded in the year 2018 that intravenous tranexamic acid reduced mortality rate due to bleeding in women with PPH, irrespective of mode of delivery. The WHO collaborator subsequently launched the update of recommendation including the administration of tranexamic acid 1 gram in PPH patients within 3 hours after birth.

Moreover, the rate of ICU admission after postpartum hemorrhage was studied revealing 15 of 21 patients (71.4%). Of which, 12 patients presented disseminated intravascular coagulation (DIC) and 2 cases death (9%). Critically-ill patients deriving from massive hemorrhage from PPH also transfusion-related acute lungs injury (TRALI), congestive heart failure, acute kidney injury and multiorgan failure.

In this study, we emphasize in patients underwent cesarean delivery with PPH (intraoperative estimated blood loss > 1,000 ml). The primary purpose is to identify the maternal outcomes after PPH. The highlighted outcome is the anesthetic management including rate of blood transfusion and incidence of patient experiencing massive blood transfusion. The secondary purposes of this study are amount of blood loss, causes of PPH and other outcomes that related to PPH such as the rate of hysterectomy and postoperative outcome eg. congestive heart failure, acute kidney injury and TRALI etc. Additionally, incidence of PPH will be studied. Data collection will be made to identify the cause of PPH, anesthetic techniques that may related to the amount of hemorrhage, medical treatment for PPH and neonatal outcomes. We also aim to obtain the rate of ICU admission and revealed the factors involving the ICU admission in PPH patients underwent cesarean delivery.

The detail of outcomes of PPH in cesarean delivered patients in Siriraj hospital is scared; and it has not yet been described in the literature. Therefore, the authors aim to collected the data and analyzed the outcomes associated with PPH, in order to report in the literatures as well as improving the anesthetic management of intraoperative PPH in our institute.

ELIGIBILITY:
Inclusion Criteria:

* Patients underwent cesarean delivery with estimated blood loss equal or more than 1,000 ml

Exclusion Criteria:

* Cesarean delivery at less than 24 weeks of gestation
* Patient chart that not contained primary outcome data eg. absent of the anesthetic record

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Female patients underwent cesarean delivery with estimated blood loss equal or more than 1,000 ml
Sampling Method: Non-Probability Sample
Enrollment: 649 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of blood transfusion | In operating theatre to 24 hour postoperatively
  Rate of blood transfusion in patients with postpartum haemorrhage
Rate of ICU admission | From 0-24 hours postoperatively
  Patients with postpartum haemorrhage required admission in the ICU

SECONDARY OUTCOMES:
Amount of haemorrhage | In operating theatre to 24 hour postoperatively
  Amount of blood loss after delivery
Rate of hysterectomy | In operating theatre to 24 hour postoperatively
  Rate of hysterectomy after postpartum hemorrhage
Anesthetic technique | In operating theatre to 24 hour postoperatively
  General anesthesia with endotracheal tube or regional anesthesia
Rate of blood component administration | In operating theatre to 24 hour postoperatively
  Rate of patients receiving FFP, cryoprecipitate or platelets
Rate of Tranexamic acid administration | In operating theatre to 24 hour postoperatively
  Rate of patients receiving Tranexamic acid
Causes of postpartum hemorrhage | In operating theatre to 24 hour postoperatively
  Identify causes of postpartum hemorrhage
Factor associated ICU admission | In operating theatre to 24 hour postoperatively
  Factor associated ICU admission after cesarean delivery with postpartum hemorrhage
Rate of complications after postpartum haemorrhage | 0-30 days postoperatively
  Rate of complications after postpartum haemorrhage eg. prolong intubation, congestive heart failure, acute kidney injury, transfusion-related acute lungs injury (TRALI)
Maternal mortality rate | 0-30 days postoperatively
  Report rate of maternal death
Neonatal outcomes | At 1 and 5 minutes after delivery
  Neonatal Apgar score

CONTACTS AND LOCATIONS:
Overall Officials: Patchareya Nivatpumin, M.D., Principal Investigator — Mahidol University
Locations (1):
- Faculty of Medicine Siriraj Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Nivatpumin P, Nithi-Uthai J, Lertbunnaphong T, Sukcharoen N, Soponsiripakdee T, Yonphan P. Perioperative outcomes and causes of postpartum hemorrhage in patients undergoing cesarean delivery in Thailand: A comprehensive retrospective study. PLoS One. 2024 Apr 16;19(4):e0300620. doi: 10.1371/journal.pone.0300620. eCollection 2024. PMID 38626161
- [Result] Nivatpumin P, Nithiuthai J, Lertbunnaphong T. The impact of the WOMAN trial on local clinical practice in Thailand. J Anesth. 2025 Oct;39(5):828-830. doi: 10.1007/s00540-025-03518-6. Epub 2025 Jun 18. PMID 40533618